CLINICAL TRIAL: NCT00204984
Title: The Effect of Aortic Impedance on Myocardial Relaxation
Brief Title: Heart and Blood Pressure Study: The Effect of Aortic Impedance on Myocardial Relaxation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-2004-0382; K23 AGO01022
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: High Blood Pressure
Keywords: arterial stiffness; echocardiography; nesiritide
MeSH Terms: conditions — Hypertension | interventions — Hydralazine

INTERVENTIONS:
Drug: oral hydralazine and intravenous nesiritide — vasodilators

SUMMARY:
Does dilation of blood vessels (vasodilation), which decreases aortic stiffness, have a greater effect on heart myocardium relaxation (diastole) than vasodilation which affects mean pressure equally without improving aortic stiffness?

DETAILED DESCRIPTION:
60 subjects, 30 with hypertension and 30 without will attend two visits to the GCRC. At each visit, pulsatile hemodynamics (by using tonometry-a non-invasive means to obtain arterial pressure tracings) and Doppler tissue imaging relaxation velocity (a measurement of myocardial relaxation obtained by echocardiography) data will be collected before and after administration of vasodilator medication. At the first visit, each patient will receive an oral dose of the vasodilator hydralazine (does not effect aortic stiffness), and at the second visit each patient will receive intravenous nesiritide (does effect aortic stiffness). The relationship between timing of the reflected pulse wave and myocardial relaxation velocity will be studied at baseline and following administration of each vasodilator to determine if changing aortic stiffness has an impact on myocardial relaxation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over the age of 65

Exclusion Criteria:

* Have known or suspected coronary artery disease
* Have known or suspected left ventricular dysfunction
* Have significant valvular, infiltrative, pericardial, or congenital heart disease
* Have a resting systolic blood pressure < 100 mmHg
* Have had an adverse reaction to nesiritide or hydralazine
* Have a serum creatinine > 2 mg/dl at Visit 1

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-05; Primary Completion 2006-12-20 (Actual); Study Completion 2006-12-20 (Actual)

PRIMARY OUTCOMES:
heart myocardium relaxation (diastole) | before and after administration of vasodilator medication

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Sweitzer, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Result] Sweitzer NK, Hetzel SJ, Skalski J, Velez M, Eggleston K, Mitchell GF. Left ventricular responses to acute changes in late systolic pressure augmentation in older adults. Am J Hypertens. 2013 Jul;26(7):866-71. doi: 10.1093/ajh/hpt043. Epub 2013 Mar 28. PMID 23537892